CLINICAL TRIAL: NCT01653496
Title: Phase II Study Evaluating the Compliance to the Enhanced Recovery After Surgery (ERAS) Program in Patients Undergoing Gastrectomy for Gastric Carcinoma
Brief Title: Compliance to ERAS After Gastric Surgery
Acronym: ERAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chonnam National University Hospital (Other)
Responsible Party: Principal Investigator, Young Kyu Park, Professor, Department of Gastroenterologic Surgery, Chonnam National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNUHGES-001
Record Dates: First submitted 2012-07-13; First posted 2012-07-31 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Stomach Neoplasms
Keywords: Gastric cancer; Perioperative care; Enhanced recovery after surgery; Multimodal rehabilitation; Fast track surgery; Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Enhanced recovery after surgery (Experimental): Patients who receive ERAS program after gastric cancer surgery
  Interventions: Procedure: Enhanced recovery after surgery

INTERVENTIONS:
Procedure: Enhanced recovery after surgery — The main 18 elements of ERAS program included are described in detail in the brief summary of the study

SUMMARY:
The purpose of this study is to prospectively evaluate the overall compliance to the enhanced recovery after surgery (ERAS) program in patients undergoing gastric cancer surgery.

DETAILED DESCRIPTION:
The feasibility and effectiveness of ERAS program for various major surgical procedures have been well studies in the literature. However, ERAS program has not been widely accepted for patients undergoing gastric cancer surgery because of the paucity of evidence about its feasibility and efficacy. In this study, we developed ERAS program for gastric cancer surgery, based on the systemic review about perioperative cares. The main elements of ERAS program includes: 1preoperative patient education, 2)no preoperative bowel preparation, 3) provision of normal diet until the night before surgery, 4)carbohydrate rich drink 2 hrs before surgery, 5)epidural anesthesia for pain control, 6) local wound anesthetic infiltration for pain control, 7)no routine abdominal drain, 8)no naso-gastric tube insertion, 9)intraoperative antibiotics, 10)thromboprophylaxis using intermittent pneumatic compression device, 11)intraoperative normothermia using warm air blanket, 12)low oxygen supply during immediate postoperative period, 13)restrictive postoperative fluid administration, 14)early postoperative oral diet, 15)early active ambulation, 16)early removal of the urinary catheter, 17)patient education before discharge, and 18)hospital discharge based on discharge criteria.

The aim of study is to evaluate the compliance to these main elements of ERAS program in patients undergoing gastric cancer surgery.

Previously reported data about ERAS program for colon surgery reported overall compliance as about 65%. Considering that this is a single center study, we expected overall compliance rate of 70%. Therefore, the sample size of 173 patients was calculated based on this expected compliance rate, with permitted error of 95% confidence interval of 14%.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are to undergo gastric cancer surgery
* ASA score < 3
* ECOG performance status 0-1
* Adequate hepatic, renal, and hematologic function
* Written informed consent

Exclusion Criteria:

* Previous abdominal operation history
* Concommitant other organ malignant disease
* Preoperative chemotherapy or radiation therapy
* Concommitant other organ resection during surgery
* Emergency operation due to bleeding or perforation
* Active underlying medical illness
* Pregnancy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2012-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Overall compliance to the ERAS program | 90 days
  Patient's compliance to the 18 main elements of ERAS program

SECONDARY OUTCOMES:
Morbidity | 90 days
  Postoperative complications means any complications occured within 90 days after operation, and will be assessed based on the predefined definition and severity of postoperative complication of our institution.
Hospital stay | 90 days
  The length of hospital stay means the duration from the operation until hospital discharge.
Mortality | 90 days
  Any death related to surgery within 90 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kyu Park, MD, PhD, Principal Investigator — Chonnam National University Hospital, Korea
Locations (1):
- Chonnam Nationl University Hwasun Hospital, Hwasun-gun, Jeollanam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jung MR, Ryu SY, Park YK, Jeong O. Compliance with an Enhanced Recovery After a Surgery Program for Patients Undergoing Gastrectomy for Gastric Carcinoma: A Phase 2 Study. Ann Surg Oncol. 2018 Aug;25(8):2366-2373. doi: 10.1245/s10434-018-6524-4. Epub 2018 May 22. PMID 29789971